CLINICAL TRIAL: NCT07263308
Title: Albumin for Patients With Acute Large Vessel Occlusive Stroke Undergoing Endovascular Therapy -2
Acronym: ARISE-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor of Neurology, Xuanwu Hospital, Capital Medical University, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARISE-2
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Acute Ischemic Stroke
Keywords: Albumin; Acute Large Vessel Occlusive Stroke; Acute Ischemic Stroke; Endovascular Therapy; China
MeSH Terms: conditions — Ischemic Stroke | interventions — Albumins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Albumin combined with endovascular treatment group (Experimental): Albumin combined with recommended endovascular treatment will be applied.
  Interventions: Drug: Albumin; Procedure: Endovascular treatment
- Endovascular treatment group (Active Comparator): Recommended endovascular treatment will be applied.
  Interventions: Procedure: Endovascular treatment

INTERVENTIONS:
Drug: Albumin — 25% human albumin at a dose of 0.5g/kg (maximum dose 37.5g) should be administered intravenously. On the second, third, and fourth days, 25% human albumin at a dose of 0.5g/kg (maximum dose 37.5g) should be administered daily.
  Arms: Albumin combined with endovascular treatment group
Procedure: Endovascular treatment — Best endovascular treatment.

SUMMARY:
This study is a prospective, multicenter, open-label, randomized controlled clinical trial. The investigators will apply albumin to the reperfusion treatment of patients with acute ischemic stroke in the anterior circulation. This study aims to verify the efficacy and safety of albumin combined with endovascular treatment in patients with anterior circulation acute ischemic stroke.

DETAILED DESCRIPTION:
This study investigates the application of albumin in reperfusion therapy for patients with acute ischemic stroke in the anterior circulation. Patients who met all inclusion criteria and none of the exclusion criteria will be randomly assigned in a 1:1 ratio to either the Albumin combined with Endovascular Therapy group or the Endovascular Therapy group. All subjects in both groups received acute stroke treatment and secondary prevention therapy according to current American stroke guidelines, aside from our intervention. At baseline, subjects underwent non-contrast cranial computed tomography (CT) or magnetic resonance angiography (MRA) to identify the occlusion site and presence of hemorrhage; relevant laboratory tests and mRS, NIHSS, and ASPECTS scores were also completed. Furthermore, vital signs were recorded. A 90-day post-randomization telephone follow-up was conducted to assess patients using several quality of life scales.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years;
2. Acute ischemic stroke with indications for endovascular treatment within 24 hours of onset;
3. Anterior circulation acute ischemic stroke, with acute occlusion of the responsible vessel located in the intracranial segment of the internal carotid artery, or the M1 or M2 segment of the middle cerebral artery;
4. National Institute of Health Stroke Scale (NIHSS) score >=6;
5. Alberta Stroke Program Early CT Score (ASPECTS) >=3 points;
6. Modified Rankin Scale (mRS) score ≤1 before onset of the disease;
7. Written informed consent provided by the patients or their legal relatives.

Exclusion Criteria:

1. Evidence of intracranial hemorrhage (intracerebral hematoma (ICH), subarachnoid hemorrhage (SAH), epidural hemorrhage, acute or chronic subdural hematoma (SDH)) on the baseline CT or MRI scan;
2. History of congenital or acquired bleeding disorders, coagulation factor deficiency diseases, thrombocytopenic diseases, etc;
3. Anticipated difficulty in completing endovascular treatment due to vascular tortuosity;
4. Known severe allergy (more severe than skin rash) to contrast agents uncontrolled by medications;
5. Pregnancy, breastfeeding;
6. An episode or exacerbation of congestive heart failure from any cause in the past 6 months;
7. History of heart valve disease complicated by congestive heart failure within the past 6 months;
8. Cardiac surgery with thoracotomy (eg. coronary artery bypass grafting or valve replacement surgery) within the past 6 months;
9. Acute myocardial infarction in the past 6 months;
10. Signs or symptoms of acute myocardial infarction upon admission, including electrocardiographic findings;
11. Elevated serum troponin concentration upon admission (>0.1 μg/L) ;
12. Acute arrhythmia (including any tachycardia or bradycardia) with hemodynamic instability (systolic blood pressure <100 mm Hg) upon admission;
13. Acute or chronic lung diseases requiring long-term or intermittent oxygen therapy;
14. Findings on physical examination of any of the following abnormalities: (1) Jugular venous distension (jugular venous pulsation >4 cm above the sternal angle); (2) Resting tachycardia due to congestive heart failure (heart rate > 100 per/min); (3) Third heart sound; (4) Abnormal hepatic jugular venous reflux; (5) Pitting edema of the lower extremities attributable to congestive heart failure or without apparent cause; (6) Rales in both lungs; (7) Or evidence of pulmonary edema, pleural effusion, or pulmonary vascular redistribution on chest X-ray;
15. Severe chronic anemia (hemoglobin < 75 g/L);
16. Known recent or current serum creatinine exceeding 1.5 times the upper limit of normal, or estimated glomerular filtration rate (eGFR) < 60 mL/min;
17. Refractory hypertension that is difficult to control by medication (defined as systolic blood pressure > 220 mmHg, or diastolic blood pressure > 110 mmHg);
18. Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) is greater than 1.5 times the upper limit of the normal value.
19. History of albumin allergy or known allergy to albumin;
20. Patients with severe mental disorders or dementia who are unable to cooperate in completing informed consent and follow-up content;
21. The expected survival time is less than 90 days (such as comorbidity with malignant tumor or severe systemic diseases etc.);
22. Patients who have participated in other interventional clinical studies within 30 days before randomization or are currently participating in other interventional clinical studies.
23. The investigator believes that the subject has other conditions making it unsuitable for participating in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1192 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2027-06-20 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with functional independence at 90 days (mRS 0-2) | 90 days

SECONDARY OUTCOMES:
Distribution of mRS scores at 90 days | 90 days
Proportion of patients with mRS score 0-1 at 90 days | 90 days
24h National Institutes of Health Stroke Scale (NIHSS) | 24 hours
  The NIHSS ranges from 0 to 42, with higher scores indicating worse outcomes.
National Institutes of Health Stroke Scale (NIHSS) at 7 days | 7 days
  The NIHSS ranges from 0 to 42, with higher scores indicating worse outcomes.
EuroQol Five-Dimension Five-Level Questionnaire (EQ-5D-5L) at 90 days | 90 days
  The EQ-5D-5L includes 5 dimensions: mobility, self-care, usual activities,pain/discomfort, and anxiety/depression. Each dimension has 5 levels: 1= no problems, 2= slight problems, 3= moderate problems, 4= severe problems, and 5= extreme problems. Higher scoresindicating worse quality of life.
Proportion of Barthel Index (BI) ≥95 at 90 days | 90 days

OTHER OUTCOMES:
The incidence of symptomatic intracerebral hemorrhage | 7 days
The incidence of newly onset atrial fibrillation within 7 days | 7 days
The incidence rate of newly onset pulmonary edema or congestive heart failure within 7 days | 7 days
All-cause mortality rate at 90 days | 90 days

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Taihe County Hospital of Traditional Chinese Medicine, Fuyang, Anhui
  - Si County People's Hospital, Suzhou, Anhui
  - Xuanwu Hospital，Capital Medical University, Beijing, Beijing Municipality
  - Shanghai General Hospital Jiujuan Hospital, Jiuquan, Gansu
  - Gansu Provincial Hospital, Lanzhou, Gansu
  - Jixi People's Hospital, Jixi, Heilongjiang
  - Ningling County People's Hospital, Shangqiu, Henan
  - The First Affiliated Hospital of Xinxiang Medical University, Weihui, Henan
  - The First Affiliated Hospital of Henan University of Chinese Medicine, Zhengzhou, Henan
  - Zhongmou County People's Hospital, Zhengzhou, Henan
  - Rizhao Hospital of Traditional Chinese Medicine, Rizhao, Shandong
  - Laizhou People's Hospital, Yantai, Shandong

IPD SHARING:
Plan to Share IPD: Undecided